CLINICAL TRIAL: NCT03503747
Title: Investigating Genetic Risk for Type 1 Diabetes
Acronym: INGR1D
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: OVG 2017/09
Record Dates: First submitted 2018-01-30; First posted 2018-04-20 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases
Keywords: type 1 diabetes; Infants; INGR1D
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to determine the percentage of children with genetic markers putting them at increased risk of developing type 1 diabetes, and to offer the opportunity for these children to be enrolled into a phase II b primary prevention trial.

DETAILED DESCRIPTION:
This is a population screening study to undertake (with prospective consent) additional testing of the newborn screening blood to identify children at increased genetic risk of type 1 diabetes. This study will enrol newborn babies whose mothers have given consent to additional testing for the newborn blood screening (routinely performed when the baby is approximately 5 days old).

Women will be approached by research staff in the second or third trimester of pregnancy (≥18 weeks gestation) when attending for antenatal care. At this point, the study will be discussed with the woman and if interested a patient information sheet will be provided as well as the opportunity to ask questions. If they agree to participate, a qualified member of the research team will take written informed consent. This consent will allow a) completion of a questionnaire and b) prospective consent to use the surplus neonatal screening blood sample for genetic testing.

The punch from the blood sample will analysed for the child's risk of type 1 diabetes. If found to be at high risk (>10%) they will be contacted by a member of the clinical study team to discuss the results and invite them to participate in a phase II prevention trial.

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian of participant is willing and able to give informed consent for participation in the study.
* Participant has provided blood for the newborn screening blood test, with sufficient sample remaining after routine testing.

Exclusion Criteria:

* Parent/legal guardian unwilling or unable to give written informed consent to participate in the study
* Unable to understand written or verbal English which would preclude them from understanding the study

Ages: 0 Months to 4 Months | Sex: All
Age Groups: Child
Study Population: The study will include all infants where the mother has consented to the additional screening test being performed.
Sampling Method: Probability Sample
Enrollment: 15640 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Quantification of the number of participants with high-risk genetic markers for the development of type 1 diabetes. | February 2021
  The number of children with a greater than 10% (high) risk of developing type 1 diabetes will be quantified, based on risk scores derived from SNPs that show the presence of HLA DR3, HLA DR4, and HLA DQ8 alleles as well as SNPs from HLA class I and non-HLA type 1 diabetes susceptibility genes, and from HLA class II protective alleles.

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, United Kingdom

REFERENCES:
- See also: Related Info — http://www.gppad.org